CLINICAL TRIAL: NCT05565495
Title: The Effects of ECMO on the Pharmacokinetics of Hydromorphone
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Xiaobo Yang, MD (Other)
Responsible Party: Sponsor-Investigator, Xiaobo Yang, MD, Clinical Professor, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Organization: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PKHM20210920
Record Dates: First submitted 2022-09-13; First posted 2022-10-04 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Extracorporeal Membrane Oxygenation
Keywords: Extracorporeal Membrane Oxygenation; Pharmacokinetics; Hydromorphone
MeSH Terms: interventions — Hydromorphone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hydromorphone (Experimental): Hydromorphone was administered intravenously at a rate of 0.03 mg/kg/h for 72 h for analgesia. Blood samples were collected before administration and at different time points after administration, and the content of hydromorphone and hydromorphone-3-glucuronide (the main metabolite) was detected by quantitative liquid chromatography tandem mass spectrometry. And then a population pharmacokinetic model of hydromorphone in patients under ECMO was established.
  Interventions: Drug: Hydromorphone

INTERVENTIONS:
Drug: Hydromorphone — Hydromorphone was administered intravenously at a rate of 0.03 mg/kg/h for 72 h for analgesia. Blood samples were collected before administration and at different time points after administration, and the contents of hydromorphone and hydromorphone-3-glucuronide (main metabolite) were detected by quantitative liquid chromatography tandem mass spectrometry, and then A population pharmacokinetic model of hydromorphone in patients under ECMO was established.

SUMMARY:
The purpose of this study was to establish a population pharmacokinetic (PPK) model of hydromorphone in patients under ECMO, and to recommend a dosing regimen when the target effective concentration was reached.

DETAILED DESCRIPTION:
A population pharmacokinetic (PPK) model of hydromorphone in patients under ECMO was established. The patients were given hydromorphone 0.03mg/kg/h by continuous intravenous infusion for 72 hours for analgesia. Blood samples were collected at different time points before and after administration, and quantitative liquid chromatography tandem mass spectrometry was used to detect hydromorphone and its main metabolite, hydromorphone-3-glucuronide.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 80;
* Using hydromorphone for pain relief;
* Using ECMO for more than 96h

Exclusion Criteria:

* Allergic to hydromorphone;
* Use of CRRT during ECMO;
* Liver function Child-Pugh B, C grade;
* Pregnancy;
* Intestinal obstruction;
* Refused to sign the informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Volume of distribution of hydromorphone and hydromorphone-3-glucuronide in patients on ECMO | Within 4 days
  Quantitative liquid chromatography-tandem mass spectrometry was used to detect the contents of hydromorphone and hydromorphone -3- glucuronide in blood samples at various time points, so as to obtain the pharmacokinetics of continuous intravenous infusion of hydromorphone for 72 hours during ECMO.

SECONDARY OUTCOMES:
Clearance of hydromorphone and hydromorphone-3-glucuronide in patients on ECMO | Within 4 days
  Clearance of hydromorphone and hydromorphone-3-glucuronide in patients on ECMO

CONTACTS AND LOCATIONS:
Locations (1):
- Wuhan Union Hospital, Wuhan, Hubei, China